CLINICAL TRIAL: NCT06493032
Title: The Use of Body Surface Gastric Mapping in Assessing the Clinical Success of G-POEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mohammad Al-Haddad, Principal Investigator, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20972
Record Dates: First submitted 2024-05-24; First posted 2024-07-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: enrolling 20 participants who are being referred for G-POEM procedure into this study for a baseline alimetry and then again at 3-6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Body Surface Gastric Mapping (Experimental)
  Interventions: Device: Gastric Alimetry System

INTERVENTIONS:
Device: Gastric Alimetry System — medical device that uses a large sheet of electrodes to assess gastric motility
  Other Names: Body Surface Gastric Mapping; BSMG; Electrogastrography System

SUMMARY:
The purpose of this study is to investigate whether or not the investigators can utilize Body Surface Gastric Mapping to determine who would best benefit to receive G-POEM procedure and how Body Surface Gastric Mapping can be utilized with patients who have gastroparesis symptoms. the investigators may also be able to find more ways how Body Surface Gastric Mapping testing can benefit patients with gastroparesis and/or G-POEM procedure.

DETAILED DESCRIPTION:
The aim of this protocol is to build on the investigators currently approved study to evaluate the outcomes and predictors of success of Gastric peroral endoscopic myotomy (G-POEM). The investigators plan to incorporate BSGM in determining the treatment success after G-POEM in patients with refractory gastroparesis and potentially identify a phenotype of gastroparesis patients who may respond more favorably to G-POEM based on their baseline BSGM profile. The currently approved G-POEM study (IRB #1708840627 and ClinicalTrials.gov ID NCT04434781) at our center tracks patients' symptoms and quality of life at baseline and post G-POEM. the investigators plan to supplement the existing study by adding BSGM variables. Although the investigators have specific outcomes identified, the investigators would like to stress that this is a pilot study that will serve to identify patterns and trends that could be studied further in the future using larger cohorts of patients.

The investigators' primary objective is to evaluate the safety and feasibility BSGM in refractory gastroparesis patients undergoing G-POEM.

the investigators will also investigate whether changes in BSGM measures correlate with changes in symptoms and quality of life.

Additionally, the investigators' aim to compare the diagnostic performance of BSGM, and gastric emptying scans as depicted on scintigraphy.

The investigators' primary aim is to assess the feasibility and safety of in gastroparesis patients undergoing G-POEM. Clinical success is defined as improvement in GCSI by 1 point or more compared to baseline.

The investigators will report four spectral metrics, each profiling distinct features of gastric function:

* Body Surface Gastric Mapping Rhythm IndexTM (GA-RI) - a measure of gastric rhythm stability.
* Principal Gastric Frequency - the frequency associated with stable, persistent gastric activity as defined by GA-RI.
* BMI-adjusted amplitude.
* Fed: Fasted Amplitude Ratio (ff-AR).

Although not directly related to this outcome, the investigators will continue our symptom analysis (as has been previously done under the existing G-POEM protocol) that includes both the pattern and severity of individual symptoms, such as vomiting, reflux, and belching. The investigators will continue to assess patient quality of life using standardized questionnaires (SF-36) at baseline and 3 months post-G-POEM as is currently done with the existing protocol.

This is an addition to an existing study protocol. The study will involve patients with refractory gastroparesis (proven on a 4-hour solid-phase gastric emptying scan, along with limited or no response (or intolerance) to at least 3 months of lifestyle adjustments, dietary modifications, and medications) who will undergo G-POEM. BSGM will be used to assess gastric motility before and after the procedure. This design allows for the collection of data at multiple time points to assess changes in BSGM phenotypes, gastroparesis symptoms, and other relevant variables over time.

The study team will enroll 20 participants who will undergo BSGM at baseline prior to G-POEM procedure and then again 3-6 months after G-POEM. The study team plan to contact participants prior to their standard of care clinic visit to ensure participants meet eligibility criteria. The study team will also explain the study over the phone using the telephone script that has been approved (Appendix 1). If they are interested in the study, the study team will schedule them for BSGM and go over prep instructions. Once the participant arrives in clinic, teh study team will consent in-person.

ELIGIBILITY:
Inclusion Criteria:

* • Patients clinically eligible for G-Poem at our center.

Exclusion Criteria:

* • Pregnant or breast-feeding

  * Patients with gastroparesis due to spinal cord injuries due to difficulties in conducting the BSGM. Of note, we rarely see gastroparesis in this context.
  * Inability to perform BSGM: history of severe skin allergies or sensitivity to cosmetics or lotions; chronically damaged or vulnerable epigastric skin (fragile skin, wounds, inflammation); patients unable to remain in a relaxed reclined position for the test duration.
  * Patients with abdominal drains or tubes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Body Surface Gastric Mapping Rhythm IndexTM (GA-RI) | Baseline, 3 months,6 months, up to 5 hours.
  A measure of the concentration of amplitude in the gastric frequency band over time (between 0 and 1), which characterizes the rhythmic stability of the recorded gastric activity; also adjusted for BMI.
Principal Gastric Frequency | Baseline, 3 months,6 months, up to 5 hours.
  Characterizes the frequency associated with stable, persistent gastric activity as defined by GA-R
BMI-Adjusted Amplitude (μV) | Baseline, 3 months,6 months, up to 5 hours.
  characterizes the strength of the recorded gastric activity as an average of the whole-test amplitude, adjusted for BMI
Fed: Fasted Amplitude Ratio (ff-AR) | Baseline, 3 months,6 months, up to 5 hours.
  characterizes the responsiveness to a meal stimulus, which is calculated as a ratio of the maximal 1-h average postprandial amplitude to the amplitude in the preprandial period.
SF-36 | Baseline, 3 months,6 months, up to 5 hours.
  a set of generic, coherent, and easily administered quality-of-life measures

SECONDARY OUTCOMES:
Body surface gastric mapping (BSMG) | Baseline, 3 months,6 months, up to 5 hours.
  enables accurate cutaneous gastric bioelectrical recording and provides valuable insights into the pathophysiology of gastric dysmotility in addition to gastric emptying measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Al-Haddad, MD, Principal Investigator — Indiana Unversity/Indiana University Health
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No